CLINICAL TRIAL: NCT05150184
Title: Isolation and Characterization of Fecal/Oral/Skin/Nasal/Throat Microbial Species From a Diverse Cohort of Healthy Adults
Brief Title: Isolation and Characterization of Multiple Microbial Species From Diverse Healthy Adults
Acronym: IsoMic
Status: Completed | Type: Observational
Sponsor: Danisco (Industry)
Collaborators: Reprocell Inc (Unknown); Serologix (Unknown)
Responsible Party: Sponsor
Other Study IDs: NH10009
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Human Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults, various ethnicities: Non-interventional
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — observational study, thus no different arm/groups

SUMMARY:
Isolation and characterization of fecal/oral/skin/nasal/throat microbial species from a diverse cohort of healthy adults.

DETAILED DESCRIPTION:
This study aims at isolation and characterizing microbial species from the diverse cohort for future development as next generation probiotics and includes the characterization of the human fecal/oral/skin/nasal and throat microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, informed consent to participate in the study
2. Agreement to comply with the protocol and study restrictions
3. Healthy females and males of age 18 to 50 years (inclusive)
4. Participants recognize themselves as white or American Indian or Alaska Native or Asian or Black / African American or Native Hawaiian or Other Pacific Islander or Hispanic and Latinos or Multiracial. Participant numbers are limited to a maximum of 10 (males and females) from each group.
5. Participants consume > 4 portions of fruits and vegetables per day and who agree to maintain their usual dietary habits, their usual exercise habits, hygienic habits and their lifestyle in general throughout the trial period
6. Females of child-bearing potential who agree to use medically approved methods of birth control
7. Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study
8. BMI between 18.5-25.

Exclusion Criteria:

1. Participation in a clinical trial with an investigational product or drug within 60 days prior to screening.
2. Likeliness to be noncompliant with the protocol, or to be unsuitable to the study as judged by the study staff for any reason.
3. Planned major changes in life style (i.e. diet, dieting, exercise level, travelling).
4. History of diagnosed eating disorder (anorexia, bulimia).
5. Consumption of fast food > 3 times/week. Where fast food is referred to high carbohydrate and fat rich diet.
6. History of drug (> 2 times per week) during last 2 years or alcohol abuse (> 08 portions per week for females and 15 portions/week for males, or >3 portions/day) during the last 3 months.
7. Pregnant or breastfeeding women; women planning to become pregnant during the study.
8. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may affect the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness, coronary heart disease/cardiovascular disease or artificial heart valve, HIV, STD, AIDS, hepatitis and autoimmune diseases e.g. MS-disease, thyroid diseases)
9. Use of prescription anti-obesity drugs, temporary or irregular medication for diabetes, dyslipidemia or hypertension, non-steroidal anti-inflammatory drugs, corticosteroids, or equivalent immunomodulatory drugs, immunosuppression or ongoing therapy causing immunosuppression and ongoing or recent (last 3 months) antibiotic treatment.
10. Diagnosed or suspected organic gastrointestinal disease (e.g. colitis, Crohn's disease, celiac disease, recurrent diverticulitis) or non-organic disease (e.g. IBS), or functional constipation, during the last year.
11. Colonoscopy within 3 months before screening
12. Colon cleansing within 3 months before screening.
13. Gastrointestinal infection within 6 months before screening
14. Active or recent (last 3 months) participation in a weight loss program including weight change (increase or loss) of 3 kg during the past three months. History of bariatric surgery.
15. History of gingivitis, periodontitis, or any oral disease during last 6 months.
16. History of smoking or tobacco use in any form and/or electronic cigarette during the last 6 months.
17. History of skin diseases (e.g. atopic dermatitis (Eczema), hives, dermatitis, psoriasis, or rashes) during the last 6 months.
18. History of SARS CoV-2 infection.
19. Participants under administrative or legal supervision.
20. Other reasons that, in the opinion of the Investigator, make the participant unsuitable for enrollment

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy donors of various ethnicities, within normal BMI range.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Analysis of microbiomes from various body sites | within 2 weeks of collection
  Analysis of microbiomes from various body sites

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A Lehman, PhD, Principal Investigator — Reprocell
Locations (1):
- Reprocell, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided as of now